CLINICAL TRIAL: NCT02189681
Title: Comparison of Conventional Landmark Guided Midline (Group C) Versus Pre-procedural Ultrasound Guided Paramedian at L5S1 (Group P) Technique for Spinal Anaesthesia
Brief Title: Landmark Guided Midline Versus Pre-procedural Ultrasound Guided Paramedian at L5S1 for Spinal Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Karthikeyan Kallidaikurichi Srinivasan, Specialist Registrar,Anaesthetics,Cork University Hospital, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: L5S1 study
Record Dates: First submitted 2014-07-05; First posted 2014-07-14 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Anaesthesia
Keywords: spinal anaesthesia; ultrasound; paramedian
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group C (Active Comparator): Patients in this group underwent Conventional landmark guided midline spinal anaesthesia.
  Interventions: Procedure: Conventional landmark guided midline spinal anaesthesia; Device: spinal anaesthesia
- Group P (Experimental): This group had pre-procedure ultrasound guided L5S1 paramedian spinal anaesthesia performed
  Interventions: Procedure: pre-procedure ultrasound guided L5S1 paramedian spinal; Device: spinal anaesthesia

INTERVENTIONS:
Procedure: Conventional landmark guided midline spinal anaesthesia — Spinal anaesthesia was administered based on conventional landmark based midline approach.
  Arms: Group C
Procedure: pre-procedure ultrasound guided L5S1 paramedian spinal — In group P, a portable ultrasound unit was used for initial pre-procedural marking. The L5 S1 interspinous space with best image of the anterior complex (ligamentum flavum dura complex- LFD) and posterior complex (posterior longitudinal ligament- PLL) was obtained. At this selected interspace, and with the probe positioned to obtain the clearest ultrasound image, a skin marker was used to mark the midpoint of the long border of the probe and the midpoints of the short borders of the probe . At the same horizontal level as the midpoint of the long border of the probe, the midpoint of the line drawn between the two short border midpoints of the probe was used as paramedian insertion point for the spinal needle.Spinal anaesthesia is then administered based on these landmarks.
  Arms: Group P
Device: spinal anaesthesia — Spinal anaesthesia is administered with appropriate spinal needle

SUMMARY:
Spinal anesthesia is widely performed using a surface landmark based 'blind' technique. Multiple passes and attempts while administering spinal anesthesia are associated with a greater incidence of post dural-puncture headache, paraesthesia and spinal hematoma.

Real time and pre-procedural neuraxial ultrasound techniques have been used to improve the success rate of spinal anesthesia. The use of real time ultrasound-guided spinal anesthesia has to date been limited to case series and case reports.Its use may be limited by the requirement for wide bore needles and the technical difficulties associated with simultaneous ultrasound scanning and needle advancement. The use of pre-procedural ultrasound has been shown to increase the first pass success rate for spinal anesthesia only in patients with difficult surface anatomic landmarks. No technique has been shown to improve the success rate of dural puncture when applied routinely to all patients. Routine use of pre-procedure ultrasound guided paramedian approach results in 50% reduction in number of passes required for spinal anaesthetic, from a study at Cork University Hospital (awaiting publication). L5-S1 is the widest interlaminar space and provides minimal contribution to overall movement of lumbar spine.This interspinous space might still be accessible even if the patient has minimal spine flexion. We also noted that spinal needle insertion via the L5-S1 interspace was associated with the fewest passes in the pre-procedure guided ultrasound group (although non-significant).

We hypothesise that the routine use of pre-procedural ultrasound-guided paramedian spinal technique at L5S1 interspinous space will result in fewer needle passes to enter the subarachnoid space when compared to the conventional landmark based midline approach.

DETAILED DESCRIPTION:
This will be a prospective, randomised, controlled study. All consented patients scheduled to undergo elective total knee or total hip arthroplasty under spinal anesthesia will be included in the study. A written informed consent will be obtained from all patients participating in the study. Patients with contraindications to spinal anesthesia (allergy to local anesthetic, coagulopathy, local infection and indeterminate neurological disease) will be excluded from the study.

The patients will be randomised using random number generating software (Research Randomizer Version 4.0 ) to undergo either conventional landmark-guided spinal anesthesia (Group C) or pre-procedural ultrasound-guided paramedian L5S1 spinal (Group P). Group allocation will be concealed by enclosing the codes in a sealed opaque envelope and will be seen by the attending anesthesiologist immediately before performing the procedure. Patients will be blinded as to their allocated study group.

In both groups, spinal anesthesia will be performed by one of three consultant anesthesiologists (FL, PL, GI), each having performed more than 75 neuraxial ultrasound scans prior to the study. On arrival to the anesthesia induction room baseline monitoring (non-invasive blood pressure, pulse oximetry and 3 lead ECG) and intravenous access will be established. The patients will be then positioned sitting on a level trolley with feet resting on a foot rest. They will be given a pillow to hug and requested to maintain an arched back posture with an assistant holding the patient to aid positioning.

In group C, the anesthesiologist will palpate the landmarks after positioning and graded the ease of palpation on a 4 point scale (easy, moderate, difficult or impossible) as described in previous studies.10 Strict asepsis will be followed throughout the procedure with anesthesiologist scrubbed prior to procedure, wearing mask and sterile gloves. The skin will be prepped with 2% Chlorhexidine (Chloraprep 3 ml applicator, CareFusion Corporation, San Diego, CA 92130,USA) following which 2-5 ml of 1% lidocaine will be used to infiltrate the skin. The anesthesiologist performing the spinal technique will be allowed to choose the appropriate needle length ( 90 or 119 mm 25 G Whitacre needle, Becton, Dickinson and Company, Franklin Lakes, New Jersey, 07417-1880, USA), gauge (25 or 22G), depth and angle of insertion. Hyperbaric bupivacaine will be used in both groups. After completion of spinal anesthetic injection, and positioning the patient in lateral decubitus, ultrasound will be used to identify the interspinous level at which the injection will be administered.

In group P, a portable ultrasound unit with a curved 2-5 MHz probe will be used for initial pre-procedural marking. A paramedian sagittal oblique view of the neuraxis will be obtained and the sacrum will be identified, following which the interlaminar space between L5 and S1 will be noted. At this interspace with the probe positioned to obtain the clearest ultrasound image of the anterior complex (ligamentum flavum dura complex- LFD) and posterior complex (posterior longitudinal ligament- PLL) possible, a skin marker will be used to mark the midpoint of the long border of the probe and the midpoints of the short borders of the probe. The medial angulation of the probe will also be noted to guide the insertion of the spinal needle. At the same horizontal level as the midpoint of the long border of the probe, the midpoint of the line drawn between the two short border midpoints of the probe will be used as paramedian insertion point for the spinal needle. A transverse median (TM) view at the same level will also be obtained and the midline will be marked. This marking will be used to aid the medial angulation of the spinal needle. Both PSO and TM views would be graded as good (both LFD and PLL visible), intermediate (either LFD or PLL visible) and poor (both LFD and PLL not visible).15 Following skin marking, care will be taken to make sure that the needle entry site will be free of ultrasound gel prior to needle insertion. In group P, the anesthesiologist will not palpate the landmarks for grading until the spinal injection is complete. Spinal anesthesia will be performed in the same aseptic manner as mentioned earlier.

In both groups the anesthesiologists will be given the option to use alternative methods if unsuccessful after 3 attempts. For patients in group C another interspinous space could be used or ultrasound employed. For patients in group P a midline approach or a conventional landmark palpation technique could be used.

The outcomes will be noted by a single observer for all patients. Due to the nature of the study, the observer will not be blinded to the groups. A timer will be used to record the various time intervals. Time for identifying landmarks in group C will be defined as time from which the anesthesiologist started palpating to identify the landmarks to completion of the process as declared by the anesthesiologist. In group P it will be defined as time from which the ultrasound probe will be placed on the skin to the anesthesiologist declaring that the markings are completed. Time taken for performing spinal anesthetic will be defined as time taken from insertion of introducer needle to completion of injection. The number of passes, defined as the number of forward advancements of the spinal needle in a given interspinous space (i.e. withdrawal and redirection of spinal needle without exiting the skin) and number of spinal needle insertion attempts (defined as the number of times the spinal needle will be withdrawn from the skin and reinserted) will be noted.10 The number of passes and attempts will be recorded either until the completion of spinal anesthetic or until the anesthesiologist converts to an alternate technique.

Incidence of radicular pain, paraesthesia and blood in the spinal needle will also be noted. All patients who experienced paraesthesia or radicular pain will be followed over the next 24 hours and any patients with persistent symptoms will be further evaluated as per department protocol.

In both groups following administration of spinal anesthesia, patients will be positioned on either left or right lateral position depending on the site of surgery. After positioning and prior to administration of sedation, patients will be asked for their peri-procedural pain scores measured using an 11 point verbal rating scale (0=no pain, 10=most pain imaginable) and peri-procedural discomfort scores measured using an 11 point verbal rating measured (0= no discomfort, 10=most discomfort imaginable). Level of block (loss of cold sensation) will be noted 30 minutes after spinal anesthetic injection. Type and dose of sedation (Midazolam +/- Propofol infusion) will be left to the discretion of the anesthesiologist.

Study Outcomes The primary outcome will be the difference in number of passes between the two groups.

Secondary outcomes includes the following,

1. Number of spinal needle insertion attempts
2. Time for identifying landmarks
3. Time taken for performing spinal anesthetic
4. Level of block
5. Incidence of radicular pain, paraesthesia and blood in the spinal needle.
6. Peri-procedural pain
7. Peri-procedural discomfort score Statistics Based on our previous study with same group of consultants done here in CUH, the average number of passes in group C was 6.4 +/-8.6 (mean +/- SD). We hypothesised that by using pre-procedural paramedian spinal done at L5S1, the number of passes could be reduced to 1.5. Fourty eight patients in each group will be needed to achieve a power of 0.8 and type 1 error of <0.05. We are hoping to randomise 60 patients per group to allow for dropouts. All data will be analysed based on intention to treat. Data will be visually inspected for normality. Categorical data were analysed using the Chi-square test. Normally distributed parametric data were analysed using Students-t test (two groups) or ANOVA (more than 2 groups). A p value of less than 0.05 will be considered significant. SPSS version 20 will be used for the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* All consented patients scheduled to undergo elective total knee or total hip arthroplasty under spinal anesthesia will be included in the study.

Exclusion Criteria:

* Patients with contraindications to spinal anesthesia (allergy to local anesthetic, coagulopathy, local infection and indeterminate neurological disease) will be excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
difference in number of passes between the two groups. | 30 minutes within completion of apinal anaesthetic
  The number of passes, defined as the number of forward advancements of the spinal needle in a given interspinous space (i.e. withdrawal and redirection of spinal needle without exiting the skin)

SECONDARY OUTCOMES:
Number of spinal needle insertion attempts | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  number of spinal needle insertion attempts (defined as the number of times the spinal needle was withdrawn from the skin and reinserted) were noted
Blood in spinal needle | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  Presence of blood in spinal needle
Time for identifying landmarks | Up to 10 minutes fraom start of plapating for landmarks - Completed once anethetist declares that markings are complete
  Time for identifying landmarks in group C was defined as time from which the anesthesiologist started palpating to identify the landmarks to completion of the process as declared by the anesthesiologist. In group P it was defined as time from which the ultrasound probe was placed on the skin to the anesthesiologist declaring that the markings are completed
Time taken for performing spinal anesthetic | Up to 45 minutes from the start of insertion of spinal needled for administration of spinal anaesthetic
  defined as time taken from insertion of introducer needle to completion of injection
Incidence of radicular pain | Up to 24 hours after administration of spinal anaesthetic
  Shooting pain going down along one of the dermatomal levels in the leg
Presence of paresthesia | Up to 24 hours after administration of spinal anaesthetic
  Paresthesia along dermatomal distribution during performing spinal anaesthetic
Grading of palpated landmarks | Up to 10 minutes fraom start of plapating for landmarks - Completed once anethetist declares that markings are complete
  Anesthesiologist palpated the landmarks after positioning and graded the ease of palpation on a 4 point scale (easy, moderate, difficult or impossible)
Peri-procedural VAS scores of pain at injection site | up to 30 minutes following spinal anaesthetic injection and prior to sedation
  After positioning and prior to administration of sedation, patients were asked for their peri-procedural pain scores measured using an 11 point verbal rating scale (0=no pain, 10=most pain imaginable)
peri-procedural discomfort scores | up to 30 minutes following spinal anaesthetic injection and prior to sedation
  peri-procedural discomfort scores measured using an 11 point verbal rating measured (0= no discomfort, 10=most discomfort imaginable).
Level of block | 15 minutes after spinal anaesthetic injection
  Dermatomal level at which loss of cold sensation (ethyl chloride spray) occurs

CONTACTS AND LOCATIONS:
Overall Officials: Karthikeyan Kallidaikurichi Srinivasan, FCARCSI,MD, Principal Investigator — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork,Ireland, Cork, Ireland